CLINICAL TRIAL: NCT03398876
Title: A Single-dose and Repeated-dose, Open-label, Randomized, Cross-over Study to Assess the Nicotine Pharmacokinetics, Tolerability and Safety With A New Oral Nicotine Replacement Product in Healthy Japanese Smokers.
Brief Title: A Study to Assess the Nicotine Pharmacokinetics, Tolerability and Safety With a New Oral Nicotine Replacement Product in Healthy Japanese Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108422; 10258820TDP1001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2017-12-22; First posted 2018-01-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Nicotine Chewing Gum; Tobacco Products

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1; Treatment Sequence ABDC (Experimental): Participants will receive Treatment A (one spray of oromucosal nicotine spray [ONS]) at Visit 1, then Treatment B (2 consecutive sprays of ONS at Visit 2, then Treatment D (1 cigarette [10 puffs]) at Visit 3, followed by Treatment C (nicotine gum) at Visit 4. The visits will be separated by a period of at least 7 calendar days.
  Interventions: Drug: Oromucosal Nicotine Spray (ONS); Drug: Nicotine Gum; Other: Cigarette
- Part 1; Treatment Sequence BCAD (Experimental): Participants will receive Treatment B at Visit 1, then Treatment C at Visit 2, then Treatment A at Visit 3 followed by Treatment D at Visit 4. The visits will be separated by a period of at least 7 calendar days.
  Interventions: Drug: Oromucosal Nicotine Spray (ONS); Drug: Nicotine Gum; Other: Cigarette
- Part 1; Treatment Sequence CDBA (Experimental): Participants will receive Treatment C at Visit 1, then Treatment D at Visit 2, then Treatment B at Visit 3 followed by Treatment A at Visit 4. The visits will be separated by a period of at least 7 calendar days. The visits will be separated by a period of at least 7 calendar days.
  Interventions: Drug: Oromucosal Nicotine Spray (ONS); Drug: Nicotine Gum; Other: Cigarette
- Part 1; Treatment Sequence DACB (Experimental): Participants will receive Treatment D at Visit 1, then Treatment A at Visit 2, then Treatment C at Visit 3 followed by Treatment B at Visit 4. The visits will be separated by a period of at least 7 calendar days.
  Interventions: Drug: Oromucosal Nicotine Spray (ONS); Drug: Nicotine Gum; Other: Cigarette
- Part 2; Treatment Sequence EF (Experimental): Participants who complete Part 1 will be selected for Part 2 based on the results of genetic polymorphism test and other examinations. Selected participants will receive Treatment E (two consecutive sprays of ONS once every 30 minutes until 11.5 hours) at Visit 5, followed by Treatment F (two consecutive sprays of ONS once every 1 hour until 11 hours) at Visit 6. The visits will be separated by a period of at least 7 calendar days.
  Interventions: Drug: Oromucosal Nicotine Spray (ONS)
- Part 2; Treatment Sequence FE (Experimental): Participants who complete Part 1 will be selected for Part 2 based on the results of genetic polymorphism test and other examinations. Selected participants will receive Treatment F at Visit 5 followed by Treatment E at Visit 6. The visits will be separated by a period of at least 7 calendar days.
  Interventions: Drug: Oromucosal Nicotine Spray (ONS)

INTERVENTIONS:
Drug: Oromucosal Nicotine Spray (ONS) — Participants will receive oral dose of oromucosal nicotine spray (ONS).
Drug: Nicotine Gum — Participants will chew nicotine gum for 30 minutes.
  Arms: Part 1; Treatment Sequence ABDC; Part 1; Treatment Sequence BCAD; Part 1; Treatment Sequence CDBA; Part 1; Treatment Sequence DACB
Other: Cigarette — Participants will smoke one cigarette as 10 puffs for 3 minutes.
  Arms: Part 1; Treatment Sequence ABDC; Part 1; Treatment Sequence BCAD; Part 1; Treatment Sequence CDBA; Part 1; Treatment Sequence DACB

SUMMARY:
In Part 1, the purpose of this study is to elucidate the single-dose pharmacokinetic profiles of 1 spray and 2 consecutive sprays of oromucosal nicotine spray (ONS) in comparison with those of nicotine gum and cigarette smoking in healthy Japanese smokers. In Part 2, the purpose is to evaluate the multiple-dose nicotine pharmacokinetics of ONS administered repeated-dose administration in healthy Japanese smokers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female Japanese participants between the ages of 20 and 50 years, inclusive. Health is defined as the absence of clinically relevant abnormalities identified by a detailed medical history, blood pressure, pulse rate measurements, 12-lead electrocardiogram (ECG) as well as clinical laboratory tests, as judged by the principal investigator or sub investigator.
* Smoking of at least 15 cigarettes daily during at least one year preceding inclusion
* Body Mass Index between 17.5 and 30.0 kilogram per square meter (kg/m^2) and a total body weight greater than or equal to (>=) 50.0 kg
* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study
* All women of childbearing potential, except for postmenopausal females, must have a negative urine beta-human chorionic gonadotropin (beta-hCG) at screening of Part 1 and all planned visits of Part 1 and Part 2

Exclusion Criteria:

* Evidence or history of an acute or chronic medical or psychiatric condition or allergy or laboratory abnormality, or of use of drugs that, in the judgment of the principal investigator or sub investigator, increase the risk associated with study participation or interfere with the interpretability of study results
* Females: Pregnancy, breast-feeding, premenopausal, or perimenopausal state with insufficient contraception
* Treatment with an investigational drug within 3 months preceding the first dose of study product
* Participant has donated blood or blood product or had substantial loss of blood more than 200 milliliter (mL) within 1 month before study products administration, or greater than or equal to (>=) 400 mL within 3 months for males and 4 months for females before study products administration, or participant has donated a total volume of blood in the past one year exceeding 1,200 mL for males and 800 mL for females, or participant has an intention to donate blood or blood products during the study and for at least 3 months for males and 4 months for females for blood, or at least 2 months for both genders for blood products after completion of the study
* Exclusion Criterion for Only Part 2: participants who is analyzed as cytochrome (CYP)2A6 *4/*4 by CYP2A6 genetic polymorphism test at Visit 1 of Part 1

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Baseline Corrected Plasma Nicotine Concentration (cCmax) | Predose; 2, 4, 6, 8, 10, 15, 20, 30, 45 and 60 minute (min) and 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
  cCmax is defined as the maximum baseline corrected plasma nicotine concentration (cCmax).
Part 1: Baseline Corrected Area Under the Plasma Nicotine Concentration versus (vs) Time Curve Until the Last Measurable Time Point (cAUCt) | Predose; 2, 4, 6, 8, 10, 15, 20, 30, 45 and 60 min and 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
  cAUCt is defined as the baseline corrected area under the plasma nicotine concentration-vs time curve until the last measurable time point.
Part 1: Baseline Corrected Area Under the Plasma Nicotine Concentration-vs Time Curve Extrapolated to Infinite (cAUC[infinity]) | Predose; 2, 4, 6, 8, 10, 15, 20, 30, 45 and 60 min and 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
  cAUC(infinity) is defined as the baseline corrected area under the plasma nicotine concentration-vs time curve extrapolated to infinite.
Part 1: Baseline Corrected Area Under the Plasma Nicotine Concentration-vs Time Curve until the Last Measurable Time Point (cAUCt) | Predose; 2, 4, 6, 8, 10, 15, 20, 30, 45 and 60 min and 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
  cAUCt is defined as baseline corrected area under the plasma nicotine concentration-vs time curve until the last measurable time point.
Part 2: Average Plasma Nicotine Concentration During the Last Dosing Interval/Intervals (Cav) | Predose, 2, 4, 6, 8, 10, 15, 20, 30 post last dose (last dose: Hour 11.5 for Treatment E and Hour 11 for Treatment F); 45 and 60 min post last dose for Treatment F
  Cav is defined as the average plasma nicotine concentration during the last dosing interval/intervals.
Part 2: Area Under the Plasma Nicotine Concentration-vs Time Curve During the Last Dosing Interval/Intervals (AUCtau) | Predose, 2, 4, 6, 8, 10, 15, 20, 30 post last dose (last dose: Hour 11.5 for Treatment E and Hour 11 for Treatment F); 45 and 60 min post last dose for Treatment F
  AUCtau is defined as the area under the plasma nicotine concentration-vs time curve during the last dosing interval/intervals.
Part 2: Maximum Plasma Nicotine Concentration During the Last Dosing Interval/Intervals (Cmax) | Predose, 2, 4, 6, 8, 10, 15, 20, 30 post last dose (last dose: Hour 11.5 for Treatment E and Hour 11 for Treatment F); 45 and 60 min post last dose for Treatment F
  Cmax is defined as maximum observed plasma nicotine concentration.

SECONDARY OUTCOMES:
Part 1: Area Under the Plasma Nicotine Concentration-vs Time Curve until 10 Minutes after Start of Administration [AUC10min], | Predose; 2, 4, 6, 8, 10 min postdose
  AUC10min is defined as the area under the plasma nicotine concentration-vs time curve until 10 minutes after start of administration.
Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose; 2, 4, 6, 8, 10, 15, 20, 30, 45 and 60 min and 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Part 1: Terminal Half-Life [t1/2] | Predose; 2, 4, 6, 8, 10, 15, 20, 30, 45 and 60 min and 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
  Terminal half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Part 1: Terminal Elimination Rate Constant (Lambda[z]) | Predose; 2, 4, 6, 8, 10, 15, 20, 30, 45 and 60 min and 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
  Lambda (z) is apparent terminal elimination rate constant, determined by linear regression using the terminal log-linear phase of the log transformed concentration-time curve.
Part 2: Minimum Plasma Nicotine Concentration During the Last Dosing Interval/Intervals (Cmin) | Predose, 2, 4, 6, 8, 10, 15, 20, 30 post last dose (last dose: Hour 11.5 for Treatment E and Hour 11 for Treatment F); 45 and 60 min post last dose for Treatment F
  Cmin is defined as the minimum plasma nicotine concentration during the last dosing interval/intervals.
Part 2: Peak-Trough Fluctuation [PTF] | Predose, 2, 4, 6, 8, 10, 15, 20, 30 post last dose (last dose: Hour 11.5 for Treatment E and Hour 11 for Treatment F); 45 and 60 min post last dose for Treatment F
  PTF calculated by 100*(Cmax - Cmin)/Cav will be assessed.
Part 2: Swing | Predose, 2, 4, 6, 8, 10, 15, 20, 30 post last dose (last dose: Hour 11.5 for Treatment E and Hour 11 for Treatment F); 45 and 60 min post last dose for Treatment F
  Swing will be calculated as (Cmax - Cmin)/Cmin.
Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose, 2, 4, 6, 8, 10, 15, 20, 30 post last dose (last dose: Hour 11.5 for Treatment E and Hour 11 for Treatment F); 45 and 60 min post last dose for Treatment F
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) | Up to 4 months
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Japan